CLINICAL TRIAL: NCT00674401
Title: RADAR-AF: Radiofrequency Ablation of Drivers of Atrial Fibrillation
Brief Title: Radiofrequency Ablation of Drivers of Atrial Fibrillation
Acronym: RADAR-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Felipe Atienza (Other)
Collaborators: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Responsible Party: Sponsor-Investigator, Felipe Atienza, MD, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNIC-13
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): In patients with paroxysmal atrial fibrillation: Empirical pulmonary vein antrum circumferential isolation.
  In patients with persistent atrial fibrillation: Empirical circumferential PV antrum isolation w/out roof line.
  Interventions: Procedure: Radiofrequency catheter ablation
- 2 (Active Comparator): In patients with paroxysmal atrial fibrillation: High frequency sites ablation in the LA.
  In patients with persistent atrial fibrillation: A combined approach involving pulmonary vein antrum isolation w/out roof line and high frequency sites ablation
  Interventions: Procedure: Radiofrequency catheter ablation

INTERVENTIONS:
Procedure: Radiofrequency catheter ablation — * In case of Paroxysmal AF, patients will be randomized into one of 2 in the study:
    1. Empirical pulmonary vein antrum circumferential isolation, or
    2. High frequency sites ablation in the LA
  * In case of Persistent AF, patients will be randomized into one of 2 in the study:
    1. Empirical circumferential PV antrum isolation w/out roof line, or
    2. A combined approach involving PV antrum isolation w/out roof line and high frequency sites ablation.

SUMMARY:
The purpose of this study is to assess the value of ablation of high frequency sources following circumferential pulmonary veins isolation in patients with paroxysmal and persistent atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia in clinical practice, accounts for one-third of arrhythmia hospitalizations and is associated with an increased risk of stroke, heart failure, and all-cause mortality. Moreover, there is an increasing AF prevalence due to aging of the population, a rising prevalence of chronic heart disease, and increased survival. Unfortunately, medications aimed at suppressing AF and maintaining sinus rhythm or at controlling ventricular rate are only marginally effective and may cause serious adverse effects. The limitations of pharmacologic treatment patterns have fuelled the development of new interventional strategies. Current techniques of AF ablation can achieve a 60-80% improvement in highly selected patients with medically refractory AF. However, the procedure is not without risk, is long-lasting and recurrence rates are still high. Moreover, the results in persistent AF patients are far from optimal, require the creation of extensive atrial lesions and repeated procedures. The main reason that explains the current situation is the incomplete understanding of mechanisms underlying AF maintenance despite many years of research and speculation. The incremental value of ablation of high frequency sources following circumferential PV isolation has not been assessed. There is no prospective data available as to the safety and benefit of such a combined approach in patients with paroxysmal and persistent AF. Such information would be very important in helping guide the future direction of ablative therapy for AF as well as helping to answer important questions about the role of high frequency sites in persistent AF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or older.
* Patients with paroxysmal AF symptomatic and refractory to at least one antiarrhythmic medication.
* In patients with paroxysmal AF, at least one episode of AF must have been documented by ECG or Holter within 12 months of randomization in the trial.
* Patients with persistent AF defined as a sustained episode that had been present for more than seven days without intervening spontaneous episodes of sinus rhythm and that recurred within seven days after cardioversion.
* Patients with persistent AF must be on continuous anticoagulation with warfarin (INR 2-3) for> 4 weeks prior to ablation. In patients with paroxysmal AF no continuous anticoagulation therapy with warfarin for > 4 weeks prior to ablation will be needed provided a transesophageal echocardiogram performed prior to ablation exclude the presence of thrombi or other abnormalities that discourage performing the procedure.
* Patients must be able and willing to provide written informed consent to participate in the clinical trial.

Exclusion Criteria:

* Patients with AF secondary to reversible causes.
* Patients with inadequate anticoagulation levels as defined in the inclusion criteria.
* Patients with left atrial thrombus, tumor, or another abnormality which precludes catheter introduction on TEE prior to the procedure.
* Patients with contraindications to systemic anticoagulation with heparin or coumadin.
* Patients who have previously undergone atrial fibrillation ablation, either by surgery or by percutaneous catheter.
* Patients with left atrial size > 55 mm.
* Patients who are or may potentially be pregnant.
* Patients with hyperthyroidism or hypothyroidism.
* Current enrollment in another investigational drug or device study.
* Pacemaker or Implantable Cardioverter Defibrillator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2009-01; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation at 6 months post-first ablation procedure off antiarrhythmic medications. | 6 month post first-ablation procedure
  Freedom from atrial fibrillation at 6 months post-first ablation procedure off antiarrhythmic medications in patients with either paroxysmal or persistent AF (primary analysis population)

SECONDARY OUTCOMES:
Freedom from atrial fibrillation on or off antiarrhythmic medications at 3, 6 and 12 months post-first ablation procedure. | 3, 6 and 12 month post-first ablation procedure
Freedom from atrial fibrillation and other atrial arrhythmias at 3, 6 and 12 months post-first ablation procedure | 3, 6 and 12 month post-first ablation
Need of redo procedures after 6 months | after 6 month of ablation procedure
Incidence of peri-procedural complications including stroke, PV stenosis, cardiac perforation, esophageal injury, and death | During the procedure and follow-up
Procedure duration | During the procedure
Fluoroscopy time | During the procedure
Quality of life measurements (SF-36) at baseline, 3, 6 and 12 months post-first procedure | Baseline, 3, 6 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Atienza, MD, Study Director — Hospital General Universitario Gregorio Marañon
Locations (11):
- Spain (11):
  - Hospital Juan Canalejo, A Coruña, A Coruña
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Hospital de Basurto, Bilbao, Bilbao
  - Clínica San Sebastian, Bilbao, Bilbao
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Grupo Hospital de Madrid, Madrid, Madrid
  - Hospital Virgen de las Nieves, Granada
  - Hospital Virgen de la Salud, Toledo

REFERENCES:
- [Derived] Atienza F, Almendral J, Ormaetxe JM, Moya A, Martinez-Alday JD, Hernandez-Madrid A, Castellanos E, Arribas F, Arias MA, Tercedor L, Peinado R, Arcocha MF, Ortiz M, Martinez-Alzamora N, Arenal A, Fernandez-Aviles F, Jalife J; RADAR-AF Investigators. Comparison of radiofrequency catheter ablation of drivers and circumferential pulmonary vein isolation in atrial fibrillation: a noninferiority randomized multicenter RADAR-AF trial. J Am Coll Cardiol. 2014 Dec 16;64(23):2455-67. doi: 10.1016/j.jacc.2014.09.053. PMID 25500229